CLINICAL TRIAL: NCT06562855
Title: Gene Expression-methylation Profiling
Brief Title: Tension-Type Headache Gene Expression and Methylation
Acronym: TTH
Status: Available | Type: Expanded Access
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Şenay Görücü Yılmaz, Prof. Dr., University of Gaziantep
Other Study IDs: GaziantepUniversity
Record Dates: First submitted 2024-05-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Tension-Type Headache, Unspecified, Intractable
Keywords: Tension-Type Headache; Gene expression; Gene methylation
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Genetic: Peripheral blood sampling

SUMMARY:
Tension-type headache (TTH) refers to pain radiating from the forehead to the back of the head as a bilateral band. It often occurs without warning and spreads to the neck muscles. Patients describe it as tension, pressure, or dull pain. It is usually triggered by stress. The complexity of the processes is the biggest difficulty in diagnosing and treating TTH. Although there are genetic connections, there are no single responsible genes.

DETAILED DESCRIPTION:
130 TTH patients and 117 healthy controls were included in the study. Serum markers of the patients were measured. WNT5A, responsible for the Wnt-B catenin signaling pathway, and its receptor FZD3 were examined in the pathogenesis of TTH. Expression changes and methylation profiles of genes were obtained. Genetic and serum parameters were compared. Diagnostic powers were determined by ROC analyses.

ELIGIBILITY:
Inclusion Criteria:

* (ICHD)-3 criteria
* Male and female
* 17-82 years
* not diagnosed with tension-type or other primary headaches

Exclusion Criteria:

* Tension-type headache not diagnosed
* below 16 ages
* pregnant woman
* subdural hematoma
* intracranial mass

Ages: 17 Years to 82 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziantep University Şahinbey Research and Application Hospital, Gaziantep, Şehitkamil
  - Medicine, Gaziantep, Şehitkamil